CLINICAL TRIAL: NCT03216356
Title: Effect of D-cycloserine on a Short Imagery Rescripting Intervention for Subclinical PTSD
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Boston University Charles River Campus (Other)
Collaborators: James S McDonnell Foundation (Other)
Responsible Party: Principal Investigator, Stefan G. Hofmann, Professor of Psychology, Boston University Charles River Campus
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 4114
Record Dates: First submitted 2016-10-18; First posted 2017-07-13 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Cycloserine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- CBT + ImRs + DCS pill (Experimental): The experimental arm involves cognitive-behavioral therapy, imagery rescripting techniques and d-cycloserine medication (pill).
  Interventions: Behavioral: CBT + ImRs; Drug: D-Cycloserine
- CBT + ImRs + placebo (Active Comparator): The active comparator arm involves cognitive behavioral therapy, imagery rescripting techniques and placebo medication (pill).
  Interventions: Behavioral: CBT + ImRs; Drug: Placebo
- CBT + I.E. + study pill (Active Comparator): The placebo comparator involves cognitive behavioral therapy, imaginal exposure and study pill (DCS or placebo)
  Interventions: Behavioral: CBT + I.E.; Drug: Study Pill

INTERVENTIONS:
Behavioral: CBT + ImRs — Cognitive Behavioral Therapy with Imagery Rescripting
  Other Names: Experimental Group
  Arms: CBT + ImRs + DCS pill; CBT + ImRs + placebo
Behavioral: CBT + I.E. — Cognitive Behavioral Therapy with Imagery Exposure
  Other Names: Active Comparison Group
  Arms: CBT + I.E. + study pill
Drug: D-Cycloserine — 250 mg DCS (derived from Seromycin 250 mg capsules)
  Other Names: Experimental Group
  Arms: CBT + ImRs + DCS pill
Drug: Placebo — polyethylene glycol 3350 powder
  Other Names: Active Comparison Group; Placebo Comparison Group
  Arms: CBT + ImRs + placebo
Drug: Study Pill — 250 mg DCS (derived from Seromycin 250 mg capsules) or polyethylene glycol 3350 powder
  Arms: CBT + I.E. + study pill

SUMMARY:
This study aims to investigate the utility of d-cycloserine (DCS) for enhancing the effect of a novel psychosocial intervention, imagery rescripting (ImRs), in adults with mild to moderate PTSD symptoms after experiencing a traumatic event such as sexual or physical assault, serious accident, etc. Participants will receive 4 sessions of either cognitive behavioral therapy with imagery rescripting or cognitive behavioral therapy with imaginal exposure and will receive study medication (DCS or Pill placebo) prior to Session 2 and Session 3.

DETAILED DESCRIPTION:
The primary aim of this proof-of-concept-study is to investigate the utility of d-cycloserine (DCS; a partial N-methyl-D-aspartate receptor agonist) for enhancing the effect of a novel psychosocial intervention, imagery rescripting (ImRs).

ImRs is a therapeutic technique that has shown positive outcomes for people suffering from PTSD and as an adjunct to CBT for PTSD. Patients are asked to recall their memory of a specific traumatic experience, and then to imagine an intervention that changes the course and outcome of the event to produce a more satisfying result. It is hypothesized that reconsolidation of the trauma memory is the mechanism of ImRs. DCS augments exposure therapy but also appears to enhance reconsolidation of memory. We hypothesize that DCS will enhance the effect of ImRs by incorporating safety cues into the trauma memory.

Sixty adults with PTSD symptoms due to a traumatic event at least three months prior to intake will receive 4 sessions of either: CBT + ImRs, or CBT + imaginal exposure (IE). In sessions 2 and 3, participants will be randomized to receive either DCS or placebo (PLA).

We hypothesize that DCS + ImRs sessions will enhance treatment outcome by facilitating reconsolidation of the trauma memories incorporating new safety cues. We also hypothesize that ImRs + PLA will provide equal or better outcomes as the IE + PLA condition.

The primary outcome measure will be improvements in PTSD symptoms, as assessed at baseline, post-treatment and at 1-month follow-up. Secondary outcome measures will be self-report questionnaires assessing depression symptoms, general psychological complaints, sleep quality, quality of life, and PTSD cognitions.

ELIGIBILITY:
Inclusion Criteria:

* Adult outpatients ≥ 18 years of age, who have experienced a traumatic event such as sexual assault, physical assualt, a serious accident, or other event where they feared for their life or their safety, at least 3 months prior to intake, with a primary subclinical psychiatric diagnosis of post-traumatic stress disorder (PTSD) as measured by the CAPS-5 (structured clinical interview to assess for PTSD according to the DSM-5). Eligible participants will have a CAPS-5 score of mild or moderate.
* Physical examination and laboratory findings within normal limits, as determined by the study nurse.
* Willingness and ability to participate in the informed consent process and comply with the requirements of the study protocol.
* Potential subjects must have sufficient command of the English language.

Exclusion Criteria:

* A lifetime history of bipolar disorder, schizophrenia, psychosis, delusional disorders or organic brain syndrome; past history of reported or current seizures; use of Isoniazid (a particular antibiotic); cognitive dysfunction that can interfere with capacity to engage in therapy;
* A history of substance or alcohol dependence (other than nicotine) in the last 6 months (or otherwise unable to commit to refraining from alcohol use during the acute period of study participation). The acute period of study participation is defined as during their visit and 24 hours before and after their visit.
* Patients with significant suicidal ideation or who have enacted suicidal behaviors within 6 months prior to intake will be excluded from study participation and referred for appropriate clinical intervention.
* Patients cannot be taking psychotropic medication during the study period. They have to be off psychotropic medication for three weeks.
* Participating in ongoing exposure-based psychotherapy for PTSD or psychodynamic therapy focusing on exploring specific, dynamic causes of the traumatic symptomatology and providing management skills. General supportive therapy initiated > 3 months prior to study is acceptable.
* Significant personality dysfunction likely to interfere with study participation. For example, overly aggressive behavior or disruptive behavior that might jeopardize safety of the staff or impairs providing the treatment.
* Serious medical illness or instability for which hospitalization may be likely within the next year. For example, if people are currently in a treatment for cancer, or people that are waiting for organ donation. This decision would be determined by our medical staff during the eligibility screen.
* Patients with a current or past history of epilepsy or seizures.
* Patients who have experienced any cardiac event. Patients with clinically significant abnormalities in vital signs (e.g., systolic blood pressure >150 mm Hg or diastolic blood pressure >100 mm Hg) at screening will be excluded from further study participation and referred for appropriate clinical management.
* Pregnant women, lactating women, women who are breastfeeding and women of childbearing potential who are not using medically accepted forms of contraception (e.g., IUD, oral contraceptives, or implanted progesterone rods stabilized for at least 3 months).
* Patients with a history of head trauma causing loss of consciousness, or ongoing cognitive impairment.
* Patients who experienced multiple events of interpersonal trauma prior to the age of 14.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-09; Primary Completion 2023-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
The Clinician-Administered PTSD Scale (CAPS) | Change from baseline to 4 weeks (post-treatment)
  The CAPS is a semi-structured interview that assesses PTSD symptom severity. It will also be administered at 1-week and 4-week follow up (see secondary outcomes)

SECONDARY OUTCOMES:
PTSD Checklist for DSM-5 (PCL-5) | Change from baseline to 4 weeks (post-treatment), 5 weeks (1-week follow-up) and 9 weeks (1- month follow-up)
  The PCL-5 is a self-reported measure of PTSD symptom severity. It will also be administered every session during treatment (weeks
Depression, Anxiety and Stress Scale (DASS-21) | Change from baseline to 4 weeks (post-treatment), 5 weeks (1-week follow-up) and 9 weeks (1- month follow-up)
  The DASS is a self-reported measure of depression, anxiety and stress. It will also be administered before every therapy session.
Posttraumatic Cognitions Inventory (PTCI) | Change from baseline to 4 weeks (post-treatment), 5 weeks (1-week follow-up) and 9 weeks (1- month follow-up)
  The PTCI measures negative cognitions about the self, the world and self-blame related to trauma. It will also be administered at every therapy session.
Pittsburgh Sleep Quality Index (PSQI) | Change from baseline to 4 weeks (post-treatment), 5 weeks (1-week follow-up) and 9 weeks (1-month follow-up)
  The PSQI measures various domains of sleep quality over the past month
Quality of Life Enjoyment and Satisfaction Questionnaire | Change from baseline to 4 weeks (post-treatment), 5 weeks (1-week follow-up) and 9 weeks (1-month follow-up)
  The Q-LES-Q measures various domains of quality of life and life satisfaction
The Clinician-Administered PTSD Scale (CAPS) at follow-up | Changes from baseline to 5 weeks (1-week follow-up) and 9 weeks (1- month follow-up)
  The CAPS is a semi-structured interview that assesses PTSD symptom severity.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph K Carpenter, M.A., Study Chair — Boston University; Megan Pinaire, B.S., Study Chair — Boston Universtiy
Locations (1):
- Center for Anxiety and Related Disorders at Boston University, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Arntz A, Weertman A. Treatment of childhood memories: theory and practice. Behav Res Ther. 1999 Aug;37(8):715-40. doi: 10.1016/s0005-7967(98)00173-9. PMID 10452174
- [Background] Lee JL, Milton AL, Everitt BJ. Reconsolidation and extinction of conditioned fear: inhibition and potentiation. J Neurosci. 2006 Sep 27;26(39):10051-6. doi: 10.1523/JNEUROSCI.2466-06.2006. PMID 17005868
- [Background] Arntz A, Tiesema M, Kindt M. Treatment of PTSD: a comparison of imaginal exposure with and without imagery rescripting. J Behav Ther Exp Psychiatry. 2007 Dec;38(4):345-70. doi: 10.1016/j.jbtep.2007.10.006. Epub 2007 Oct 26. PMID 18005935
- [Background] Hofmann SG, Smits JA, Rosenfield D, Simon N, Otto MW, Meuret AE, Marques L, Fang A, Tart C, Pollack MH. D-Cycloserine as an augmentation strategy with cognitive-behavioral therapy for social anxiety disorder. Am J Psychiatry. 2013 Jul;170(7):751-8. doi: 10.1176/appi.ajp.2013.12070974. PMID 23599046
- [Background] Litz BT, Salters-Pedneault K, Steenkamp MM, Hermos JA, Bryant RA, Otto MW, Hofmann SG. A randomized placebo-controlled trial of D-cycloserine and exposure therapy for posttraumatic stress disorder. J Psychiatr Res. 2012 Sep;46(9):1184-90. doi: 10.1016/j.jpsychires.2012.05.006. Epub 2012 Jun 12. PMID 22694905
- [Background] Arntz A, Sofi D, van Breukelen G. Imagery Rescripting as treatment for complicated PTSD in refugees: a multiple baseline case series study. Behav Res Ther. 2013 Jun;51(6):274-83. doi: 10.1016/j.brat.2013.02.009. Epub 2013 Mar 6. PMID 23524061